CLINICAL TRIAL: NCT00004219
Title: A Study to Investigate the Efficacy and Tolerability of Two Dose Levels of Lerisetron Compared With Granisetron in Patients Receiving Radiotherapy for Stage I Seminoma
Brief Title: Lerisetron Compared With Granisetron in Preventing Nausea and Vomiting in Men Being Treated With Radiation Therapy for Stage I Seminoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Simbec Research (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: SIMBEC-RD526/21494; CDR0000067456 (Registry Identifier: PDQ (Physician Data Query)); EU-99027
Record Dates: First submitted 2000-01-28; First posted 2004-08-09 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2007-06

CONDITIONS: Nausea and Vomiting; Testicular Germ Cell Tumor
Keywords: nausea and vomiting; stage I malignant testicular germ cell tumor; testicular seminoma
MeSH Terms: conditions — Nausea; Vomiting; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma | interventions — Granisetron; lerisetron; Radiotherapy

INTERVENTIONS:
Drug: granisetron hydrochloride
Drug: lerisetron
Radiation: radiation therapy

SUMMARY:
RATIONALE: Antiemetic drugs may help to reduce or prevent nausea and vomiting in patients treated with radiation therapy. It is not yet known whether lerisetron is more effective than granisetron in preventing nausea and vomiting.

PURPOSE: Randomized phase III trial to compare the effectiveness of lerisetron with that of granisetron in preventing nausea and vomiting in men who are being treated with radiation therapy for stage I seminoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy and safety of lerisetron versus granisetron hydrochloride in the prevention of radiotherapy induced nausea and vomiting in men with stage I testicular seminoma.

OUTLINE: This is a randomized, double blind, parallel, multicenter study. Patients are randomized to one of three treatment arms. Arm I: Patients receive oral lerisetron with an oral placebo once daily for 14 days. Arm II: Patients receive oral lerisetron once daily for 14 days. Arm III: Patients receive oral granisetron hydrochloride once daily for 14 days. At 1-2 hours following antiemetics, all patients undergo concurrent daily radiotherapy for at least 10 out of 14 days. Patients are followed daily for 10 days.

PROJECTED ACCRUAL: A total of 150 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of stage I seminoma No clinical evidence of brain metastases

PATIENT CHARACTERISTICS: Age: 18 to 70 Sex: Male Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No significant hepatic impairment Renal: No significant renal impairment Other: No known hypersensitivity to serotonin antagonists No prior anticipatory emesis No communication impairments (e.g., language problem, poor mental development, or impaired cerebral function) that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No concurrent corticosteroids except topical 1% hydrocortisone or equivalent Radiotherapy: No prior radiotherapy Surgery: Not specified Other: At least 48 hours since prior antiemetics No other concurrent antiemetics

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David P. Dearnaley, MD, FRCP, FRCR, Study Chair — Royal Marsden NHS Foundation Trust